CLINICAL TRIAL: NCT01096446
Title: Tolerance of Higher Infusion Rates of Intravenous Fat Emulsions in Extremely Low Birthweight Infants During the First Week of Life
Brief Title: Intravenous Fat Emulsions and Premature Infants
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: To many infants in the experimental group developed hypertriglyceridemia
Sponsor: OSF Healthcare System (Other)
Responsible Party: Principal Investigator, Kamlesh Macwan, Neonatalogist, OSF Healthcare System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OSF-118
Record Dates: First submitted 2010-03-30; First posted 2010-03-31 (Estimated); Results first posted 2014-11-20 (Estimated); Last update posted 2014-11-20 (Estimated); Status verified 2014-11

CONDITIONS: Hypertriglyceridemia; Hyperglycemia
MeSH Terms: conditions — Hypertriglyceridemia; Hyperglycemia | interventions — Fat Emulsions, Intravenous

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Higher Infusion (Experimental): Infants randomized into the experimental group will receive 2 gm/kg/day of Intravenous Fat Emulsions (IVFE) on their first day of total parenteral nutrition (TPN). The IVFE will be increased by 0.5 gm/kg/day daily until a goal reached of 3 gm/kg/day of IVFE in the TPN.
  Interventions: Drug: Intravenous Fat Emulsions
- Standard Infusion (Other): Infants randomized into the control group will receive 0.5 gm/kg/day of Intravenous Fat Emulsions (IVFE) on their first day of total parenteral nutrition (TPN). The IVFE will be increased by 0.5 gm/kg/day daily until a goal reached of 3 gm/kg/day of IVFE in the TPN.
  Interventions: Drug: Intravenous Fat Emulsions

INTERVENTIONS:
Drug: Intravenous Fat Emulsions — Control Group: 0.5 grams/kg/day Experimental Group: 2 grams/kg/day
  Other Names: Intralipid 20%

SUMMARY:
The purpose of this study is to study the tolerances of Extremely Low Birthweight Infants who are born at less than 750 grams who are started at a higher infusion rate of intravenous lipid emulsions (2 gm/kg/day). These infants will be compared with a control group who are at the standard lipid emulsion infusion rate (0.5 gm/kg/day).

hypothesis:

A. Objectives of this project.

Null Hypothesis: There will not be a significant difference for Extremely Low Birth Weight Infants (ELBW) <750 grams being able to tolerate a higher infusion rate of Intravenous Fat Emulsions (IVFE) within the first days of life (days 1-7) as evidenced by maintenance of a serum triglyceride level of 200 mg/dl or less.

Alternative Hypothesis: There will be a significant difference (p<0.05) for Extremely Low Birth Weight Infants (ELBW) <750 grams being able to tolerate a higher infusion rate of Intravenous Fat Emulsions (IVFE) within the first days of life (days 1-7) as evidenced by maintenance of a serum triglyceride level of 200 mg/dl or less.

DETAILED DESCRIPTION:
ELBW infants will be randomized into either the control group or the experimental group.

The control group will receive standardized care which consists of receiving TPN within 24 to 36 hours of life. The control group will be given the standardized dosage of IVFE starting at 0.5 grams/kg/day in the TPN and have IVFE advanced daily by 0.5 grams/kg/day until a goal rate of 3 grams/kg/day is achieved. The experimental group will receive TPN within 24 to 36 hours of life. For these infants, IVFE will begin at 2 grams/kg/day. For the experimental group, Intralipid will be increased by 0.5 grams/kg/day until a goal rate of 3 grams/kg/day is achieved.

An informed consent form (Appendix A), to be signed by the parent or guardian, will be obtained for all infants before they are enrolled into this study. Assent waiver is requested on the study participants because they are infants.

All infants enrolled in this study will have their laboratory data monitored at least daily during the first week of life. A baseline triglyceride will be drawn prior to beginning TPN to verify that their serum triglyceride levels are <200 gm/dl. This will include a daily lipid profile panel used to evaluate the serum triglyceride levels and the tolerance of the two different IVFE infusion rates. Lipid tolerance will be defined as infants having a serum triglyceride levels at < 200 mg/dl. Lipid intolerance will be defined as infants having a serum triglyceride of 201 mg/dl or greater. If lipid intolerance occurs, IVFE will be decreased by the following standard of care:

Serum Triglycerides Levels Changes Intralipid in TPN by:

150-200 mg/dl Keep at current IVFE order 201-249 mg/dl decrease by 1 grams/kg/day 250-299 mg/dl decrease by 1.5 gram/kg/day 300 mg/dl or greater Reduce Intralipid to 0.5 grams/kg/day to prevent essential fatty acid deficiency (EFAD). If hypertriglyceridemia persists (300 mg/dlor greater) over 24 hours keep IVFE at 0.5 gm/kg/day to prevent EFAD.

The total caloric intake will be calculated and collected daily for both groups. The calorie intake will be specified as total kilocalories per kilogram (kcal/kg/day). The goal calorie intake for both groups will be 90 kcal/kg/day. The kcal/kg index will be calculated by a Registered Dietitian, who is assigned to the Neonatal Intensive Care Unit.

All collected data will be presented as a mean +/- SD. The statistical significance will be defined by a p value < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* All infants will be recruited who are admitted to the Neonatal Intensive Care Unit at Children's Hospital of Illinois.
* A total of 70 ELBW infants classified as Appropriate for Gestational Age (AGA) and who are between 500 grams to 750 grams in weight at birth.

Thirty-five infants will be randomized into the control group and thirty-five infants will be randomized into the experimental group.

Exclusion Criteria:

* Have a baseline triglyceridemia above 200 mg/dl prior to beginning the study.
* Who are classified as Small for Gestational Age (SGA)
* Who have any congenial anomalies, and/or,
* Who are septic

Ages: 1 Day to 2 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 19 (Actual)
Dates: Start 2008-04; Primary Completion 2010-05 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kamlesh S Macwan, MD, Principal Investigator — University of Illinois College of Medicine at Peoria
Locations (1):
- Children's Hospital of Illinois at OSF Saint Francis Medical Center, Peoria, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Infants with a birthweight < 750 grams were recruited from April 2008 through March 2010 at the neonatal intensive care unit at at the Children's Hospital of Illinois at OSF Saint Francis Medical Center Peoria, IL.
Pre-assignment Details: Thirty-five infants were deemed eligible for the study of which 13 infants were excluded due to one parent refused, 12 other infants were started on TPN prior to obtaining informed consent.
Period: Overall Study
Arm/Group | Higher Infusion | Standard Infusion
Started | 12 | 10
Completed | 9 (One infant was SGA; one infant had a congenital anomaly; and one discontinued medical management) | 10
Not Completed | 3 | 0
Not completed — Death | 1 | 0
Not completed — Protocol Violation | 2 | 0

BASELINE CHARACTERISTICS:
Population: Twelve infants were randomized into the experimental arm and 10 infants were randomized into the control arm.
Groups:
- Standard Infusion: Infants randomized into the experimental group will receive 0.5 gm/kg/day of Intravenous Fat Emulsions (IVFE) on their first day of total parenteral nutrition (TPN). The IVFE will be increased by 0.5 gm/kg/day daily until a goal reached of 3 gm/kg/day of IVFE in the TPN.
- Higher Infusion: Infants randomized into the control group will receive 2 gm/kg/day of Intravenous Fat Emulsions (IVFE) on their first day of total parenteral nutrition (TPN). The IVFE will be increased by 0.5 gm/kg/day daily until a goal reached of 3 gm/kg/day of IVFE in the TPN.
- Total: Total of all reporting groups
Arm/Group | Standard Infusion | Higher Infusion | Total
Number analyzed (Participants) | 10 | 12 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 10 | 12 | 22
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: weeks] — Gestational Age
  weeks | 23.7 (0.68) | 24.33 (1) | 24 (0.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 9 | 14
  Male | 5 | 3 | 8
Region of Enrollment [Number; unit: participants]
  United States | 10 | 12 | 22

OUTCOME MEASURES:

1. Primary Outcome: Number of Infants Serum Triglyceride Level Higher Than 200 mg/dl
Description: Each day the infants have a serum triglyceride level drawn to assess their tolerance of the intravenous fat emulsion being given.
Time Frame: First 7 days of life
Population: This study was ended early due to 100% of the infants in the experimental group developed hypertriglyceridemia of 200 mg/dl or greater
Measure: Number; unit: participants
Arm/Group | Higher Infusion | Standard Infusion
Number analyzed (Participants) | 9 | 10
participants | 9 | 4
Statistical Analysis 1: Comparison: Higher Infusion vs Standard Infusion; Four infants(44%)in the control group developed hypertriglyceridemia (>200 mg/dl) while 100% of the infants in the experimental group developed hypertriglyceridemia (>200 mg/dl) during the first week of life; Test type: Non-Inferiority or Equivalence — The Chi Square satistical calculation was used for analysis; p = 0.011, Chi-squared

2. Secondary Outcome: Regain Birthweight
Description: Infants in both groups weights were monitored to determine if giving higher infusions of intravenous fat emulsion helped the infants regain their birthweight sooner.
Time Frame: First 2 weeks of life
Reporting Status: Not Posted

3. Secondary Outcome: Infants Will Achieve 90 Calories/Kilogram/Day
Description: Monitored the calorie intake of infants to see which group was able to acheive 90 cal/kg/day from the total parenteral nutrition.
Time Frame: First 14 days of Life
Reporting Status: Not Posted

4. Secondary Outcome: Maintain Appropriate for Gestational Age Status at Discharge
Description: Recorded all infant's weights at discharge and plotted the anthropometric values on the Fenton Growth Charts.
Time Frame: Entire hospital stay
Reporting Status: Not Posted

5. Secondary Outcome: Initiation of Glucose
Description: Infants were monitored to see if insulin was started to control hyperglycemia.
Time Frame: First 7 days of life
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: There were no adverse events reported.
Groups:
- Serum Triglycerides: Serum triglycerides <201 mg/dl in both arms were considered to be normal. If serum triglycerides in either arm was above 201 mg/dl than the Intralipids was decreased based on the algorithm for adjusting IVFE when hypertriglyceridemia occured.
Arm/Group | Serum Triglycerides
Serious Adverse Events (participants affected / at risk) | 0/19
Other Adverse Events (participants affected / at risk) | 0/19

LIMITATIONS AND CAVEATS:
This study was terminated early because 100% of the infants in the experimental grouped developed hypertriglyceridemia (>200 gm/dl), which did not support our primary hypothesis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes